CLINICAL TRIAL: NCT03660878
Title: A Multi-Center, Double-Masked, Randomized, Parallel-Group, Vehicle-Controlled, Methodology Development Environmental Clinical Trial With Reproxalap Ophthalmic Solutions (0.25% and 0.5%) in Subjects With Seasonal Allergic Conjunctivitis
Brief Title: A Methodology Development Environmental Clinical Trial of Reproxalap in Subjects With Seasonal Allergic Conjunctivitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-AC-010
Record Dates: First submitted 2018-08-31; First posted 2018-09-07 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2018-08

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Reproxalap Ophthalmic Solution (0.25%) (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Reproxalap Ophthalmic Solution (0.5%) (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.5%)
- Vehicle Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) administered four times a day and an additional four times a day on an as needed basis.
  Arms: Reproxalap Ophthalmic Solution (0.25%)
Drug: Reproxalap Ophthalmic Solution (0.5%) — Reproxalap Ophthalmic Solution (0.5%) administered four times a day and an additional four times a day on an as needed basis.
  Arms: Reproxalap Ophthalmic Solution (0.5%)
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution administered four times a day and an additional four times a day on an as needed basis.
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
A Multi-Center, Double-Masked, Randomized, Parallel-Group, Vehicle-Controlled, Methodology Development Environmental Clinical Trial with Reproxalap Ophthalmic Solutions (0.25% and 0.5%) in Subjects with Seasonal Allergic Conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age of either gender and any race
* have a positive history of ocular allergies and a positive skin test reaction to ragweed pollen as confirmed by the allergic skin test given to the subject within 24 months of the subject's Visit 1
* have a calculated visual acuity of 0.7 logMAR or better in each eye as measured using an ETDRS chart

Exclusion Criteria:

* have known contraindications or sensitivities to the use of any of the investigational product medication or components
* have any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters (including but not limited to narrow angle glaucoma, clinically significant blepharitis, follicular conjunctivitis, iritis, pterygium, or a diagnosis of dry eye)
* have had ocular surgical intervention within three months prior to Visit 1, or during the trial, or a history of refractive surgery six months prior to Visit 1, or have systemic surgery planned during the clinical trial or within 30 days after;
* have a known history of retinal detachment, diabetic retinopathy, or active retinal disease
* have an active ocular infection (bacterial, viral or fungal), active uveitis, or positive history of an ocular herpetic infection at any visit;
* be a female who is currently pregnant, planning a pregnancy, or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-09-08 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Slade & Baker Vision, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cavanagh B, Gomes PJ, Starr CE, Nichols KK, Brady TC. Reproxalap Activity and Estimation of Clinically Relevant Thresholds for Ocular Itching and Redness in a Randomized Allergic Conjunctivitis Field Trial. Ophthalmol Ther. 2022 Aug;11(4):1449-1461. doi: 10.1007/s40123-022-00520-z. Epub 2022 May 18. PMID 35585427

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-to-treat population
Groups:
- Reproxalap Ophthalmic Solution (0.25%); Reproxalap Ophthalmic Solution (0.5%): Reproxalap administered four times daily, plus up to four more doses daily as needed, for 4 weeks
- Vehicle Ophthalmic Solution: Vehicle administered four times daily, plus up to four more doses daily as needed, for 4 weeks
Period: Overall Study
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution
Started | 18 | 17 | 17
Completed | 17 | 15 | 17
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 18 | 17 | 17 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 16 | 48
  >=65 years | 2 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 11 | 35
  Male | 5 | 6 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 11 | 30
  Not Hispanic or Latino | 8 | 8 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Black or African American | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 15 | 17 | 16 | 48
  Unknown | 0 | 0 | 0 | 0
  Not Reported | 0 | 0 | 0 | 0
  Other | 1 | 0 | 0 | 1
  Multiple | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 17 | 52
Iris Color (Right Eye) [Count of Participants; unit: Participants]
  Black | 1 | 0 | 1 | 2
  Blue | 3 | 3 | 2 | 8
  Brown | 10 | 10 | 13 | 33
  Hazel | 1 | 2 | 1 | 4
  Green | 3 | 2 | 0 | 5
  Gray | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0
Iris Color (Left Eye) [Count of Participants; unit: Participants]
  Black | 1 | 0 | 1 | 2
  Blue | 3 | 3 | 2 | 8
  Brown | 10 | 10 | 13 | 33
  Hazel | 1 | 2 | 1 | 4
  Green | 3 | 2 | 0 | 5
  Gray | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Ocular Itching Score on High Pollen Days
Description: Mean change from baseline in ocular itching score using a 0 to 4 scale (0 = least, 4 = most) was assessed on days when peak pollen counts meet or exceed the American Academy of Allergy Asthma & Immunology weed pollen scale 95th percentile (325 grains per cubic meter). The least squares mean (standard error) was derived from analysis of covariance with baseline, treatment, and day as factors.
Time Frame: Efficacy was assessed on high-pollen days over 28 days of treatment; baseline was assessed approximately one week before dosing.
Population: Intent-to-treat population and subjects with pollen count greater than 325 grains per cubic meter.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Vehicle Ophthalmic Solution | Reproxalap Ophthalmic Solution (0.5%)
Number analyzed (Participants) | 5 | 4 | 5
units on a scale | -0.65 (0.17) | 0.16 (0.18) | -0.69 (0.30)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject in the clinical trial was approximately five weeks.
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/17 | 0/17
Other Adverse Events (participants affected / at risk) | 14/18 | 16/17 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap Ophthalmic Solution (0.25%) (N=18) | Reproxalap Ophthalmic Solution (0.5%) (N=17) | Vehicle Ophthalmic Solution (N=17)
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0 — The non-ocular serious adverse event was deemed not related to study drug by the Principal Investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap Ophthalmic Solution (0.25%) (N=18) | Reproxalap Ophthalmic Solution (0.5%) (N=17) | Vehicle Ophthalmic Solution (N=17)
Skin test positive (Investigations) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1
Conjunctival disorder (Eye disorders) | 1 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0
Eye Swelling (Eye disorders) | 0 | 0 | 1
Punctate keratitis (Eye disorders) | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 1 | 0 | 0
Vitreous floaters (Nervous system disorders) | 1 | 0 | 0
Instillation site erythema (General disorders) | 0 | 1 | 0
General disorders and administration site conditions (General disorders) | 13 | 16 | 0 — Transient and self-limiting instillation site irritation that resolved in all cases. All adverse events were deemed mild by the Principal Investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT03660878/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT03660878/SAP_001.pdf